CLINICAL TRIAL: NCT05057442
Title: The Effects of Remnant-Preserving Anterior Cruciate Ligament Reconstruction on Proprioception and Functionality
Status: Completed | Type: Observational
Sponsor: Acibadem University (Other)
Collaborators: Marmara University (Other)
Responsible Party: Principal Investigator, Özgül Öztürk, Assistant Professor, Acibadem University
Other Study IDs: ATADEK 2021 / 16
Record Dates: First submitted 2021-09-16; First posted 2021-09-27 (Actual); Last update posted 2022-05-20 (Actual); Status verified 2022-05

CONDITIONS: Anterior Cruciate Ligament Rupture
MeSH Terms: conditions — Anterior Cruciate Ligament Injuries

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Anterior Cruciate Ligament Reconstruction
  Interventions: Other: Proprioception assessment, functionality assessment

INTERVENTIONS:
Other: Proprioception assessment, functionality assessment — Proprioception assessment, functionality assessment

SUMMARY:
Anterior cruciate ligament (ACL) reconstruction is a frequently performed surgical procedure to stabilize the knee joint biomechanically. At the same time, one of the goals is to improve clinical outcomes and return the patient to their daily life as early and ready as possible, as well as to sports activities. Remnant-preserving anterior cruciate ligament reconstruction is one of the reconstruction approaches that aim to achieve these goals earlier and more safely than the standard surgical procedure. However, there is no consensus in the literature regarding the effects of remnant-preserving ACL reconstruction on clinical outcomes and its superiority over the standard surgical procedure. Therefore, the aim of our study is to compare the proprioception and functionality of patients who underwent ACL reconstruction with the remnant-preserving approach, by classifying them according to stump size.

ELIGIBILITY:
Inclusion Criteria:

* Aged between 18 - 45 years,
* Anatomical single-bundle ACL reconstruction with antero-medial portal technique using hamstring autograft due to a full-thickness ACL tear,
* Endobutton technique was used for femoral fixation,
* Has not had any trauma or surgery on the non-operated knee,
* Patients with a follow-up period of at least 12 months after surgery.

Exclusion Criteria:

* Fracture of lower extremity, posterior cruciate ligament, inner and outer lateral ligament tears accompanying anterior cruciate ligament tear,
* Patients who have undergone previous surgery on the targeted knee,
* Have a revision anterior cruciate ligament reconstruction,
* Having a history of knee joint arthritis (osteoarthritis, inflammatory arthritis),
* Have a neurological disease,

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Study Population: Patients who were underwent remnant-preserving anterior cruciate ligament reconstruction
Sampling Method: Non-Probability Sample
Enrollment: 65 (Actual)
Dates: Start 2021-10-01 (Actual); Primary Completion 2022-05-05 (Actual); Study Completion 2022-05-10 (Actual)

PRIMARY OUTCOMES:
Proprioception assessment | 1 day
  Biodex® System Pro 4 (Biodex Cor. Shirley NY, USA) device will be used to evaluate the proprioception of the knee joint. The subjects will be asked to sit on the isokinetic dynamometer device with the knee joint in 90º flexion. The proprioception sense of the operated and non-operated knees will be measured at three different angles of 20º, 50º and 70º. Before the test, the procedures during the test such as knee flexion-extension, target angle and target angle recall will be assessed when eyes are open and closed. The test will be explained and actively demonstrated to all subjects before starting the assessment. During the test, the target angle will be displayed by the device and the limb will be held in this position for 10 seconds.
The Lysholm Score | 1 day
  The Lysholm Scale is used to evaluate the functionality of the knee joint, has a score between 0 and 100 points. In this scoring system, a higher score indicates a better functionality.
Single Leg Hop Test | 1 day
  Single leg forward hop test will be used to determine the functional performance level of the patient depending on the dynamic stability of the knee. The participant will be asked to stand on the leg to be tested at the starting point of the tape measure, whose toes are fixed to the floor, and to jump forward and as far as possible on the leg to be tested, along the tape measure line without losing balance. If the balance is disturbed and the foot touches the ground, the test will be repeated. There will be a one-time trial to learn the test. The test will be repeated 3 times with a 30-second rest period in between.

CONTACTS AND LOCATIONS:
Locations (1):
- Marmara University Department of Physiotherapy and Rehabilitation, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No